CLINICAL TRIAL: NCT05989022
Title: Comparison of Low-dose Spiral Breast CT With MRI in Major Indications of MRI for Breast Diagnostics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AB-CT - Advanced Breast-CT GmbH (Industry)
Collaborators: CRO Dr. med Kottmann GmbH & Co. KG (Industry); RQM+ (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ldBCT-MRI-C
Record Dates: First submitted 2023-07-25; First posted 2023-08-14 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer Diagnosis
Keywords: Breast CT
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Comparison between both modalities in single patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Imaging Breast Diagnostic (Other): Imaging breast diagnostic where patients receive both modalities MRI and B-CT to compare the resolution of the two different diagnostic devices in the same patient
  Interventions: Diagnostic Test: Injection of contrast enhancing agent Gadovist for MRI investigation; Diagnostic Test: Injection of contrast enhancing agent Imeron for B-CT investigation

INTERVENTIONS:
Diagnostic Test: Injection of contrast enhancing agent Gadovist for MRI investigation — Image enhancing contrast agent will be injected to enhance MRI resolution in breast cancer diagnosis
Diagnostic Test: Injection of contrast enhancing agent Imeron for B-CT investigation — Image enhancing contrast agent will be injected to enhance B-CT resolution in breast cancer diagnosis

SUMMARY:
Comparison between two diagnostic modalities for breast cancer diagnosis. Two different imaging systems are compared to evaluate the performance of the two systems

DETAILED DESCRIPTION:
The diagnostic quality of MRI of the breast has made this method a gold standard in the imaging of senologic lesions. Low-dose dedicated breast CT (BCT) with single photon-detection (nu:view, developed by AB-CT - Advanced Breast-CT GmbH) has emerged as a fully 3D imaging modality that uses ionizing radiation comparable to 2D mammography and has its intended use in helping with diagnosis in diagnostic breast imaging.

The investigation is designed as a prospective non-randomized intra-individual cohort procedure comparison between the imaging platforms, nu:view and MRI. Across 3 hospital-based study sites in two countries, study participants (patients who meet study criteria and have consented) sequentially receive nu:view imaging and, with a delay of up to one week (preferably on the same day), MRI imaging. At both times, patients receive contrast agent. Images generated from breasts are evaluated by three independent radiologists and their scores and interpretations are statistically evaluated. The research aim is to demonstrate non-inferiority of BCT compared with MRI in major indications of MRI for breast diagnostics.

The perceived gain in the study is to generate data on clinical performance of the BCT device nu:view and on the procedure that could be supportive of a tailored use of nu:view in patients with major indications of MRI for breast diagnostics.

ELIGIBILITY:
Inclusion Criteria:

1. Sex: female
2. Age: at least 18 years
3. Inconclusive findings in conventional imaging or preoperative staging or evaluation of therapy response in the neoadjuvant chemotherapy setting or imaging of the breast after breast-conserving therapy or finding the cause of hemorrhagic nipple discharge or prosthesis imaging or screening of women with hereditary or familial increased risk for the development of breast cancer or axillary lymph node metastasis suspected to originate from breast tissue
4. Persons able and willing to understand and sign informed consent form

Exclusion Criteria:

1. Known pregnancy or breastfeeding
2. Presence of BRCA1 or BRCA2 allele
3. Insufficient renal function (MDRD)
4. Dysfunction of the thyroid gland (TSH degradation)
5. Known allergy or intolerance against iodine-containing contrast enhancing agents or MRI contrast enhancing agents
6. Patients with paramagnetic or magnetic material inside the breast, claustrophobia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women
Enrollment: 428 (Estimated)
Dates: Start 2023-11-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of CE-BCT compared with CE-MRI in Breast Cancer diagnosis | one year
  The primary objective is to demonstrate non-inferiority of CE-BCT with CE-MRI in the BI-RADS detection at the lesion level in the diagnosis of eight indications for CE-MRI diagnosis.
  Patients with with major indications of CE-MRI will receive an additional diagnosis with CE-BCT. The images of both modalities will be compared by 3 independent raters which were randomly assigned to pseudonymized images. That rating follow the six BI-RADS Scales on lesion basis. The descriptive data will be compared according the evaluated BI-RADS scores of the raters and both modalities. For the non-inferiority test, the mean difference of lesion-wise BI-RADS scores between modalities will be used; it is expected that the mean BI-RADS values at lesion level are almost equal for both modalities.

SECONDARY OUTCOMES:
Collect data for comfort of CE-BCT and CE-MRI | one year
  The secondary objective is to collect data for comfort of CE-BCT and CE-MRI using a patient questionnaire of closed questions. The questionnaire asks in 7 categories for 1. Overall rating of the examination 2. Comfort of the device during examination 3. The feel of the operating noise of the device 4. The rating of the space provided by the device 5. The duration of the examination 6. The question if the patient would agree to have the examination again, if necessary with the device 7. After both modalities which diagnostic method would be the preference, MRI or BCT. Every question can be rated with 5 possible ratings from very good to very bad or adapted possibilities like pleasantly quit to unpleasantly loud.

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (2):
  - DRZ Die Radiologen, Regensburg, Bavaria
  - Radiologisches Institut Universitätsklinikum Erlangen, Erlangen
- Netherlands (2):
  - Stichting Martini Ziekenhuis, Groningen
  - Leiden University Medical Centre, Leiden

IPD SHARING:
Plan to Share IPD: No